CLINICAL TRIAL: NCT00995969
Title: A Randomized, Double-Blind, Placebo Controlled Phase II, Multi-Centre, Study of the Efficacy and Safety of CT 327, a Topical Cream Formulation of Pegylated K252a, When Administered Twice Daily for Eight Weeks to Patients With Mild to Moderate Psoriasis Vulgaris
Brief Title: CT 327 in the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creabilis SA (Industry)
Responsible Party: Professor Nikhil Yawalkar, Inselspital Bern
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT 327 PV 01-09
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Psoriasis
Keywords: Mild to moderate psoriasis vulgaris
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo only (Placebo Comparator): Subjects will apply placebo cream to both target lesions
  Interventions: Drug: placebo
- Active plus placebo (Active Comparator): Subjects will apply CT 327 to one target lesion and placebo to the other target lesion
  Interventions: Drug: CT 327

INTERVENTIONS:
Drug: placebo — 1.0 g (w/w) placebo cream applied to both target lesions twice daily
  Arms: Placebo only
Drug: CT 327 — 1.0 g CT 327 cream will be applied to one target lesion twice daily and 1.0 g placebo cream will be applied to the remaining target lesion twice daily
  Arms: Active plus placebo

SUMMARY:
This study will look at how safe and effective, a novel agent, CT 327 cream is in treating patients with mild to moderate psoriasis vulgaris (PV). Patients will be treated twice daily for 8 weeks on specific lesions of PV and safety and symptoms of PV will be assessed throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 71 years of age
* Able to give informed consent
* Diagnosis of mild (affecting < 3% BSA) to moderate (affecting < 10% BSA) Psoriasis Vulgaris, including, at baseline visit, two symmetrical lesions of at least 10 cm2 each

Exclusion Criteria:

* If female of childbearing potential not using an adequate and appropriate form of contraception such as oral contraceptive; intra-uterine device (IUD); contraceptive injection, implant or patch
* If female, are pregnant or lactating, or intend to become pregnant during the study period and one month thereafter
* Allergy to test drug or excipients
* Usage of topical corticosteroids or other topical treatments for PV within the last two weeks prior to study entry (including calcineurin inhibitor, topical H1 antihistamines, topical antimicrobials, other medicated topical agents) or herbal preparation to the area selected for treatment Within 4 weeks prior to study entry, have received systemic treatment for psoriasis (including systemic corticosteroids, nonsteroidals, immunosuppressants, or immunomodulating drugs, or treatment with light).
* Received treatment with systemic or locally acting medications which might counter or influence the study aim
* Presence of major medical illness requiring systemic therapy including cancers
* Clinical diagnosis of bacterial infection of the skin including impetigo and abscesses
* Any clinical relevant ECG abnormality
* Have any clinically significant abnormal clinical laboratory test results at screening
* Received any investigational drug or taking part in any clinical study within three months prior to this study
* History of drug, alcohol or other substance abuse or other factors limiting the ability to co-operate and to comply with this protocol
* Have concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug
* Have immune-compromised status (such as known human immunodeficiency virus infection)
* Have a history of malignancy, excluding basal cell carcinoma of the skin
* Have an active intercurrent infection
* Suffer from erythrodermic psoriasis, psoriasis punctata and pustular psoriasis or extended chronic stationary forms of psoriasis
* Have symptoms of a clinically significant illness that may influence the outcome of the study
* Have any reason which, in the opinion of the investigator, interferes with the ability of the subject to participate in or complete the trial, or which places the subject at undue risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Improvements from baseline on m-Psoriasis Area Severity Index Scale (m-PASI - modified to exclude area assessment): Proportion of subjects with a reduction in score of > 50% at Week 8 | 8 weeks

SECONDARY OUTCOMES:
To assess the efficacy of an 8-week treatment of CT 327 vs Placebo in terms of improvements from baseline on: Proportion of subjects with a reduction in m-PASI-score of > 75% a Week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Metrolina Medical Research, Charlotte, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, LLC, Winston-Salem, North Carolina
  - Premier Medical Group, P.C., Clarksville, Tennessee
  - East Tennessee Medical Research, Johnson City, Tennessee
- Switzerland (4):
  - University Hospital, Basel
  - Inselspital, Bern
  - Kantonsspital, Sankt Gallen
  - University Hospital, Zurich
- United Kingdom (3):
  - Synexus Midlands, Birmingham, Midlands
  - Synexus Scotland, Clydebank, Strathclyde
  - Synexus Wales, Cardiff